CLINICAL TRIAL: NCT01007877
Title: 'Study to Investigate the Effects of an Energy Drink During a 15-minute Break Versus Continued Driving on Driving Performance in the STISIM Driving Simulator'
Brief Title: Energy Drinks & Driving Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: Red Bull GmbH (Unknown)
Responsible Party: Joris C Verster, Utrecht University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 09-037
Record Dates: First submitted 2009-10-13; First posted 2009-11-04 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Driver Sleepiness
Keywords: sleepiness; driving
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No break (No Intervention)
  Interventions: Other: Red Bull Energy drink
- Placebo Energy Drink (Placebo Comparator): During a 15 minute break, subjects consume a placebo energy drink
  Interventions: Other: Red Bull Energy drink
- Red Bull Energy Drink (Experimental): during a 15 minute break, subjects consume Red Bull Energy Drink
  Interventions: Other: Red Bull Energy drink

INTERVENTIONS:
Other: Red Bull Energy drink — During a 15 minute break, subjects consume 250 ml of Red Bull® Energy Drink or placebo. Before and after the break, a 2 hour driving test is scheduled.

SUMMARY:
Rationale: Sleepiness behind the wheel is the cause of many traffic accidents. It is claimed that a 15-minute break and consuming an energy drink such as Red Bull® Energy Drink counteracts driver sleepiness.

Objective: The objective of this study is to compare driving simulator performance after (1) a 15-minute break with placebo, (2) a 15-minute break with Red Bull® Energy Drink, and (3) continued driving.

Study design: A double-blind, placebo-controlled crossover study. Study population: Healthy human volunteers, 21-35 years old.

Intervention: Each subject performs 3 test days:

1. 4 hours continued driving
2. 2 hours driving, a 15-minute break + Red Bull® Energy Drink, followed by 2 hours driving
3. 2 hours driving, a 15-minute break + placebo, followed by 2 hours driving Main study parameters/endpoints: Standard Deviation of Lateral Position (SDLP), i.e. the weaving of the car.

ELIGIBILITY:
Inclusion Criteria:

* He/she is aged between 21 and 35 years old
* BMI between 21 and 30,
* 55-85 kg body weight
* Non smoker
* Written informed consent
* Normal static binocular acuity, corrected or uncorrected
* Normal hearing
* Possession of a valid driver's license for at least 3 years
* Regular driver (> 5000 km / year)
* Be considered as reliable and mentally capable of adhering to the protocol.

Exclusion Criteria:

* Current drug use (positive urine drug screen on the presence of amphetamines (including MDMA), barbiturates, cannabinoids, benzodiazepines, cocaine, and opiates) as will be assessed by a urine drug test
* Use of psychoactive medication
* Pregnancy
* Positive alcohol breath test
* Prior enrolment in the same study
* Physical or mental illness
* Excessive alcohol use (>21 alcoholic drinks per week)
* Intake of caffeine-containing beverages under 2 or over 4 glasses per day
* Regular consumption of Energy Drinks (>1 per month)
* Shift worker (or no regular sleep pattern)
* Epworth Sleepiness Score (ESS) > 10

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP). This a measure of weaving of the car within the right traffic lane | the 2 hours of driving following the intervention

SECONDARY OUTCOMES:
Number of collisions | the 2 hours of driving following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joris Verster, PhD, Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Mets MA, Ketzer S, Blom C, van Gerven MH, van Willigenburg GM, Olivier B, Verster JC. Positive effects of Red Bull(R) Energy Drink on driving performance during prolonged driving. Psychopharmacology (Berl). 2011 Apr;214(3):737-45. doi: 10.1007/s00213-010-2078-2. Epub 2010 Nov 10. PMID 21063868